CLINICAL TRIAL: NCT04720846
Title: Assessment of a Categorized Physical Therapy Protocol for Non-arthritic Hip and Groin Pain: a Randomized Controlled Study
Brief Title: Categorized PT for Non-arthritic Hip and Groin Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2019-2120
Record Dates: First submitted 2021-01-19; First posted 2021-01-22 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-04

CONDITIONS: Hip Pain; Groin Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Active Comparator): Patients will receive standard-of-care physical therapy.
  Interventions: Other: Standard-of-care physical therapy
- Matrix-Based PT (Experimental): Patients will receive matrix-based physical therapy, in addition to standard-of-care physical therapy.
  Interventions: Other: Matrix-based physical therapy; Other: Standard-of-care physical therapy

INTERVENTIONS:
Other: Matrix-based physical therapy — Matrix-based physical therapy will be physical therapy that is based on the matrix categorization of the patient (stiff vs. mobile hips, weak vs. strong hips) and involves instructions on the amount of time that should be spent doing stretching and strengthening therapy.
  Arms: Matrix-Based PT
Other: Standard-of-care physical therapy — Physical therapy that is being conducted as standard-of-care

SUMMARY:
There is currently limited literature on a categorized physical therapy protocol for management of hip pain. Only a handful of studies have looked at the treatment of osteoarthritis of the hip with a standardized physical therapy treatment, primarily looking at manual therapy versus exercise therapy protocols. However, there are no studies observing the effect of a standardized physical therapy program on patients presenting with non-arthritic hip and groin pain. Based on the gap in the literature, this study will aim to assess the effect of matrix-based standard of care therapy in patients presenting with non-arthritic hip and groin pain.

ELIGIBILITY:
Inclusion Criteria:

* New patient presenting with non-arthritic hip impingement, hip pain, and groin pain (Tonnis 0-1)
* 18-60 years old

Exclusion Criteria:

* Arthritic hip pain (Tonnis 2+)
* <18 and >60 years old
* History of spinal fusion surgery
* History of low back pain with radicular pain
* History of hip arthroscopy
* History of inflammatory conditions, and other concurrent problems interfering with hip therapy (i.e., concurrent back/knee/foot/ankle/shoulder issues)
* Patients currently taking TNF-alpha inhibitors for inflammatory conditions
* History of prior knee osteotomy
* Non-English speakers

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2020-12-02 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
iHOT-12 (International Hip Outcome Tool-12) | Up to 6 months
  iHOT-12 is used to assess quality of life in patients with hip disorders. Scores range from 0 to 100; a higher score represents a better quality of life.

SECONDARY OUTCOMES:
NRS (numerical rating scale) pain | Up to 6 months
  NRS pain will be used to assess pain. Scores range from 0-10, with 10 representing the worst pain imaginable.
Home exercise completion | Up to 6 months
  This will be defined as the number of times patients completed their home exercises during the previous week.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Moley, MD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No